CLINICAL TRIAL: NCT02692482
Title: Effectiveness of the Use of a New Polyurethane Foam Multilayer Dressing in the Sacral Area to Prevent the Onset of Pressure Sores in the Elderly With Hip Fractures. Randomized Controlled Trial.
Brief Title: Polyurethane Foam on the Sacrum for Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22022016
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-03

CONDITIONS: Hip Fracture; Pressure Ulcer
MeSH Terms: conditions — Hip Fractures; Pressure Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- polyurethane foam (Experimental): Hydrocellular polyurethane foam multilayer dressing shaped for the sacral area
  Interventions: Device: hydrocellular polyurethane foam multilayer dressing; Procedure: standard care
- standard care (Active Comparator)
  Interventions: Procedure: standard care

INTERVENTIONS:
Device: hydrocellular polyurethane foam multilayer dressing — Application of hydrocellular polyurethane foam in the sacral region within 24 hours of admission and replaced when detaches or gets wet or dirty in addition to standard care
  Other Names: allevyn life
  Arms: polyurethane foam
Procedure: standard care — Standard care: PU risk assessment using the Braden scale within 24 hours of admission. Place patient on pressure mattress (static or alternating pressure) if Braden score <18, daily inspection of the skin in the various pressure points and moving the patient every 4 hours after surgery. Management of possible incontinence, humidity control and prevention of skin damage and rubbing/friction during postural changes as per hospital procedure.

SUMMARY:
The aim of the present study is to assess whether the application of a new hydrocellular polyurethane foam multilayer dressing shaped for the sacral area (MSP) in addition to standard care reduces the rate of pressure sores (PU) and their severity especially in the elderly population admitted for fragility Hip Fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 65 years with Hip fragility fracture without National Pressure Ulcers Advisory Panel scale (NPUAP) scale grade ≥ II PU
* Patients or legal guardians who give their consent to take part in the study

Exclusion Criteria

* Patients with known allergy to the product being tested or dermatological diseases that prevent the use of topical products
* Patients with peri-prosthetic or pathological fractures
* Patients with diaphyseal or distal femoral fractures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 359 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Polyurethane Foam | Standard Care
Started | 177 | 182
Completed | 174 | 178
Not Completed | 3 | 4
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polyurethane Foam | Standard Care | Total
Number analyzed (Participants) | 177 | 182 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.3 (7.7) | 83.2 (7.7) | 83.7 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 145 | 289
  Male | 33 | 37 | 70
Number of Participants with Neck Fracture [Count of Participants; unit: Participants] | 94 | 94 | 188
Braden score [Mean (Standard Deviation); unit: units on a scale] — The scale is composed of six subscales that reflect sensory perception, skin moisture, activity, mobility, friction and shear, and nutritional status. Each category is rated on a scale of 1 to 4, excluding the 'friction and shear' category which is rated on a 1-3 scale. This combines for a possible total of 23 points, with a higher score meaning a lower risk of developing a pressure ulcer and vice versa. The critical cut-off point at which the patient could be judged to be at risk for pressure sore formation was a Braden Scale score equal to or less than 16
  units on a scale | 15.4 (2.4) | 15.4 (2.0) | 15.4 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pressure Sores
Time Frame: On the eighth day of hospitalization or upon discharge from hospital, if that occurs before the eighth day.
Measure: Count of Participants; unit: Participants
Arm/Group | Polyurethane Foam | Standard Care
Number analyzed (Participants) | 177 | 182
Participants | 8 | 28

2. Secondary Outcome: Number of Participants With Pressure Ulcers in Other Areas (Heel, Back and Calf)
Time Frame: On the eighth day of hospitalization or upon discharge from hospital, if that occurs before the eighth day.
Measure: Count of Participants; unit: Participants
Arm/Group | Polyurethane Foam | Standard Care
Number analyzed (Participants) | 177 | 182
Participants | 7 | 7

3. Secondary Outcome: Pressure Ulcer Rate in the Sacral Area of Grade ≥ II According to the National Pressure Ulcers Advisory Panel Classification
Description: Pressure ulcer are classified and described through the use of staging systems. Staging systems describe the extent of tissue loss and the physical appearance of the injury caused by pressure and/or shear. From stage 1 (intact skin) to Stage 4 (Full-thickness skin and tissue loss).
Time Frame: On the eighth day of hospitalization or upon discharge from hospital, if that occurs before the eighth day.
Measure: Count of Participants; unit: Participants
Arm/Group | Polyurethane Foam | Standard Care
Number analyzed (Participants) | 177 | 182
Participants | 6 | 17

4. Secondary Outcome: Number of Participants With Skin Irritation/Damage Due to the Adhesive Dressing
Description: Clinical evaluation. It refers to any sort of inflammation and/or discoloration that distorts the skin's normal appearance. The skin may become scaly, bumpy, itchy, or otherwise irritated.
Time Frame: On the eighth day of hospitalization or upon discharge from hospital, if that occurs before the eighth day.
Measure: Count of Participants; unit: Participants
Arm/Group | Polyurethane Foam | Standard Care
Number analyzed (Participants) | 177 | 182
Participants | 2 | 0

ADVERSE EVENTS:
Arm/Group | Polyurethane Foam | Standard Care
All-Cause Mortality (participants affected / at risk) | 2/177 | 2/182
Serious Adverse Events (participants affected / at risk) | 0/177 | 0/182
Other Adverse Events (participants affected / at risk) | 0/177 | 0/182

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No